CLINICAL TRIAL: NCT04092894
Title: Effects of the Orexin Receptor Antagonist Suvorexant on Sleep Architecture and Delirium in the Intensive Care Unit: A Multi-Centric Randomized Controlled Trial
Brief Title: Suvorexant and Sleep/Delirium in ICU Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Professor of Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P000759
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-09

CONDITIONS: Insomnia; Sleep Fragmentation; Sleep Initiation and Maintenance Disorders; Postoperative Delirium
Keywords: Suvorexant; Sleep architecture; Delirium; Intensive care unit
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Deprivation; Emergence Delirium; Delirium | interventions — suvorexant

STUDY DESIGN:
Intervention Model Description: Randomization in a 1:1 ratio (suvorexant 20 mg versus placebo) will be stratified by duration of perioperative anesthesia and sedation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Suvorexant (Active Comparator): Suvorexant 20 mg will be administered p.o. once a day between 9:00pm and 10:00pm for 7 days starting the night after extubation in the ICU.
  Interventions: Drug: Suvorexant 20 mg
- Placebo (Placebo Comparator): Placebo will be administered p.o. once a day between 9:00pm and 10:00pm for 7 days starting the night after extubation in the ICU.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Suvorexant 20 mg — Administration of oral Suvorexant 20 mg
  Other Names: Belsomra
  Arms: Suvorexant
Drug: Placebo oral tablet — Administration of oral placebo (same non-identifiable form as active comparator)
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Investigators will evaluate the efficacy of postoperative oral suvorexant treatment on nighttime wakefulness after persistent sleep onset (WASO) among adult cardiac surgical patients recovering in the cardiac intensive care unit (ICU). The study include patients ≥ 60 years old undergoing coronary artery bypass graft surgery (CABG), with or without valve surgery (aortic or mitral). Patients will receive either oral suvorexant or placebo for 7 nights starting the night after extubation. The primary hypothesis is that suvorexant compared with placebo decreases WASO, as measured by a specialized electroencephalogram (EEG), the SedLine monitor, during the first night in the cardiac ICU. Investigators will also assess total sleep time (TST), time to sleep onset (TSO), and postoperative delirium and delirium-free days.

DETAILED DESCRIPTION:
This is a prospective, randomized, placebo-controlled, blinded study. Participants will be enrolled preoperatively. After postoperative extubation, eligible patients will be randomly allocated in a 1:1 ratio to receive either suvorexant 20 mg or placebo.

Study procedures will start on preoperative night 3 when the patient is first asked to report information about their sleep using the Richards-Campbell Sleep Questionnaire (RCSQ). Patients will complete the RCSQ every morning during the 3 days prior to surgery. The intervention (study drug) will be applied for 7 nights starting the night after postoperative extubation in the ICU. Primary and secondary outcomes will be assessed once during the night of the sleep trial in the ICU. The sleep trial will take place during the first night after extubation if the patient has been extubated before 7pm. Exploratory outcomes will be assessed from day of extubation until hospital discharge.

Suvorexant 20 mg or placebo will be administered p.o. once a day between 9:00pm and 10:00pm for a maximum of 7 days starting the night after extubation in the ICU. The study drug will be discontinued after 7 consecutive doses following extubation; or at hospital discharge (if less than 7 days after extubation); or at ICU discharge, if patient showed signs of airway obstruction during sleep or when strong inhibitors of CYP3A are co-administered; or in the event of early termination, subject withdrawal of consent, investigator withdrawal for toxicity or other reasons.

If deemed necessary by the treating clinicians, melatonin or benzodiazepine may be added for treatment of insomnia. All patients will receive usual supportive care as per the treating physicians and standard practice.

Duration of nighttime wakefulness after persistent sleep onset (WASO), total sleep time (TST), time to sleep onset (TSO) will be measured by electroencephalogram (EEG) using a Next Generation SedLine® Brain Function Monitor during the night of the sleep trial. Incidence of postoperative in-hospital delirium and increases delirium free days will be assessed using Confusion Assessment Method (CAM).

ELIGIBILITY:
Inclusion criteria:

1. Age 60 years or older
2. Undergoing elective coronary artery bypass graft surgery with or without aortic and/or mitral valve replacement, who are expected to be transferred to the ICU postoperatively

Exclusion criteria:

1. Preoperative left ventricular ejection fraction of less than 30%
2. Renal failure (creatinine >2 mg/dl or dialysis dependence)
3. Liver failure (CHILD-Pugh>4)
4. Coma (RASS<-1)
5. Signs and symptoms of delirium and agitation at time of enrollment (CAM-ICU positive)
6. Montreal Cognitive Assessment (MoCA) below 23 at time of consent
7. Psychiatric or neurologic diseases (including chronic benzodiazepine use, bipolar disorder, psychotic disorder, posttraumatic stress disorder, requirement of prophylactic psychiatric medication, evidence of acute depression on screening visit, preexisting cognitive impairment, Alzheimer disease, Parkinson's disease, medications for cognitive decline, history of recent seizures (within 1 year prior visit), alcoholism or documented history of alcohol abuse, and narcolepsy)
8. Severe sleep apnea requiring home continuous positive airway pressure treatment
9. Morbid obesity (BMI >40)
10. Known or suspected pregnancy (there are no adequate and well-controlled studies of suvorexant in pregnant women. Based on animal data, Suvorexant may cause fetal harm).
11. Patients with known hypersensitivity to study medications
12. English language limitations (Sleep assessment and delirium assessment tools are only validated in English)
13. Patients enrolled in other interventional studies which could confound the primary endpoint.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine; Balachundhar Subramaniam, Principal Investigator — Beths Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Montefiore Medical Center/Albert Einstein college of Medicine, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
The investigators intend to share de-identified individual participant data that underlie the results reported in the published article following reasonable requests to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available beginning 9 months and ending 36 months after article publication.
Access Criteria: Data will be made available to qualified scientific researchers who provide a methodologically sounds proposal following reasonable requests to the principal investigator.

REFERENCES:
- [Background] Figueroa-Ramos MI, Arroyo-Novoa CM, Lee KA, Padilla G, Puntillo KA. Sleep and delirium in ICU patients: a review of mechanisms and manifestations. Intensive Care Med. 2009 May;35(5):781-95. doi: 10.1007/s00134-009-1397-4. Epub 2009 Jan 23. PMID 19165463
- [Background] Timm FP, Zaremba S, Grabitz SD, Farhan HN, Zaremba S, Siliski E, Shin CH, Muse S, Friedrich S, Mojica JE, Kurth T, Ramachandran SK, Eikermann M. Effects of Opioids Given to Facilitate Mechanical Ventilation on Sleep Apnea After Extubation in the Intensive Care Unit. Sleep. 2018 Jan 1;41(1). doi: 10.1093/sleep/zsx191. PMID 29182729
- [Background] Herring WJ, Connor KM, Snyder E, Snavely DB, Morin CM, Lines C, Michelson D. Effects of suvorexant on the Insomnia Severity Index in patients with insomnia: analysis of pooled phase 3 data. Sleep Med. 2019 Apr;56:219-223. doi: 10.1016/j.sleep.2018.09.010. Epub 2018 Oct 2. PMID 30522875
- [Background] Herring WJ, Snyder E, Budd K, Hutzelmann J, Snavely D, Liu K, Lines C, Roth T, Michelson D. Orexin receptor antagonism for treatment of insomnia: a randomized clinical trial of suvorexant. Neurology. 2012 Dec 4;79(23):2265-74. doi: 10.1212/WNL.0b013e31827688ee. Epub 2012 Nov 28. PMID 23197752
- [Background] Michelson D, Snyder E, Paradis E, Chengan-Liu M, Snavely DB, Hutzelmann J, Walsh JK, Krystal AD, Benca RM, Cohn M, Lines C, Roth T, Herring WJ. Safety and efficacy of suvorexant during 1-year treatment of insomnia with subsequent abrupt treatment discontinuation: a phase 3 randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2014 May;13(5):461-71. doi: 10.1016/S1474-4422(14)70053-5. Epub 2014 Mar 27. PMID 24680372
- [Background] Sun H, Kennedy WP, Wilbraham D, Lewis N, Calder N, Li X, Ma J, Yee KL, Ermlich S, Mangin E, Lines C, Rosen L, Chodakewitz J, Murphy GM. Effects of suvorexant, an orexin receptor antagonist, on sleep parameters as measured by polysomnography in healthy men. Sleep. 2013 Feb 1;36(2):259-67. doi: 10.5665/sleep.2386. PMID 23372274
- [Background] Bourne RS, Minelli C, Mills GH, Kandler R. Clinical review: Sleep measurement in critical care patients: research and clinical implications. Crit Care. 2007;11(4):226. doi: 10.1186/cc5966. PMID 17764582
- [Background] Kamdar BB, Shah PA, King LM, Kho ME, Zhou X, Colantuoni E, Collop NA, Needham DM. Patient-nurse interrater reliability and agreement of the Richards-Campbell sleep questionnaire. Am J Crit Care. 2012 Jul;21(4):261-9. doi: 10.4037/ajcc2012111. PMID 22751369
- [Background] Berry RB, Brooks R, Gamaldo C, Harding SM, Lloyd RM, Quan SF, Troester MT, Vaughn BV. AASM Scoring Manual Updates for 2017 (Version 2.4). J Clin Sleep Med. 2017 May 15;13(5):665-666. doi: 10.5664/jcsm.6576. No abstract available. PMID 28416048
- [Background] Vacas S, McInrue E, Gropper MA, Maze M, Zak R, Lim E, Leung JM. The Feasibility and Utility of Continuous Sleep Monitoring in Critically Ill Patients Using a Portable Electroencephalography Monitor. Anesth Analg. 2016 Jul;123(1):206-12. doi: 10.1213/ANE.0000000000001330. PMID 27159066
- [Background] Drouot X, Roche-Campo F, Thille AW, Cabello B, Galia F, Margarit L, d'Ortho MP, Brochard L. A new classification for sleep analysis in critically ill patients. Sleep Med. 2012 Jan;13(1):7-14. doi: 10.1016/j.sleep.2011.07.012. Epub 2011 Dec 6. PMID 22153778
- [Background] Younes M, Ostrowski M, Soiferman M, Younes H, Younes M, Raneri J, Hanly P. Odds ratio product of sleep EEG as a continuous measure of sleep state. Sleep. 2015 Apr 1;38(4):641-54. doi: 10.5665/sleep.4588. PMID 25348125
- [Background] Dres M, Younes M, Rittayamai N, Kendzerska T, Telias I, Grieco DL, Pham T, Junhasavasdikul D, Chau E, Mehta S, Wilcox ME, Leung R, Drouot X, Brochard L. Sleep and Pathological Wakefulness at the Time of Liberation from Mechanical Ventilation (SLEEWE). A Prospective Multicenter Physiological Study. Am J Respir Crit Care Med. 2019 May 1;199(9):1106-1115. doi: 10.1164/rccm.201811-2119OC. PMID 30818966
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Hatta K, Kishi Y, Wada K, Takeuchi T, Ito S, Kurata A, Murakami K, Sugita M, Usui C, Nakamura H; DELIRIA-J Group. Preventive Effects of Suvorexant on Delirium: A Randomized Placebo-Controlled Trial. J Clin Psychiatry. 2017 Sep/Oct;78(8):e970-e979. doi: 10.4088/JCP.16m11194. PMID 28767209
- [Background] Tamura K, Maruyama T, Sakurai S. Preventive Effect of Suvorexant for Postoperative Delirium after Coronary Artery Bypass Grafting. Ann Thorac Cardiovasc Surg. 2019 Feb 20;25(1):26-31. doi: 10.5761/atcs.oa.18-00038. Epub 2018 Aug 9. PMID 30089761
- [Background] Herring WJ, Connor KM, Snyder E, Snavely DB, Zhang Y, Hutzelmann J, Matzura-Wolfe D, Benca RM, Krystal AD, Walsh JK, Lines C, Roth T, Michelson D. Suvorexant in Elderly Patients with Insomnia: Pooled Analyses of Data from Phase III Randomized Controlled Clinical Trials. Am J Geriatr Psychiatry. 2017 Jul;25(7):791-802. doi: 10.1016/j.jagp.2017.03.004. Epub 2017 Mar 8. PMID 28427826
- [Derived] Azimaraghi O, Hammer M, Santer P, Platzbecker K, Althoff FC, Patrocinio M, Grabitz SD, Wongtangman K, Rumyantsev S, Xu X, Schaefer MS, Fuller PM, Subramaniam B, Eikermann M. Study protocol for a randomised controlled trial evaluating the effects of the orexin receptor antagonist suvorexant on sleep architecture and delirium in the intensive care unit. BMJ Open. 2020 Jul 19;10(7):e038474. doi: 10.1136/bmjopen-2020-038474. PMID 32690536

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Suvorexant | Placebo
Started | 49 | 51
Received study drug | 47 | 47
Completed | 37 | 41
Not Completed | 12 | 10
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Discontinued EEG after randomization | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suvorexant | Placebo | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [63 to 73] | 70 [65 to 73] | 69 [64 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 37 | 39 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 29 | 25 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 17 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 33 | 34 | 67
  Unknown or Not Reported | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Nighttime Wakefulness After Persistent Sleep Onset (WASO)
Description: Nighttime wakefulness after persistent sleep onset (WASO) will be measured using a SedLine® Brain Function Monitor. WASO will be defined as the duration of wakefulness after the onset of persistent sleep in the observation period between 11:00pm (Lights-Off) to 6:00am (Lights-On) in minutes. Onset of persistent sleep will be defined as the first epoch of 10 consecutive minutes of sleep (REM or non-REM Stages 1, 2, 3 or 4) after Lights-Off. Wakefulness will be defined as any epoch of Stage 0. Sleep staging will be performed according to Rechtschaffen & Kales criteria and in accordance with AASM guidelines. The SedLine® monitor uses a symmetrical bilateral array of sensors that provides four-channel data.
Time Frame: First night after extubation between 11:00pm and 6:00am
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 37 | 41
minutes | 200.7 [112.1 to 328.4] | 184.2 [80.4 to 304.2]

2. Secondary Outcome: Total Sleep Time (TST)
Description: Total sleep time will be measured by electroencephalogram (EEG) using a Next Generation SedLine® Brain Function Monitor during the night of the sleep trial in analogy to the primary outcome.
Time Frame: First night after extubation between 11:00pm and 6:00am
Measure: Median (Inter-Quartile Range); unit: minuts
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 37 | 41
minuts | 224 [112 to 379] | 253 [68 to 420]

3. Other Pre Specified Outcome: Time to Sleep Onset (TSO)
Description: Sleep onset latency will be measured by electroencephalogram (EEG) using a Next Generation SedLine® Brain Function Monitor during the night of the sleep trial in analogy to the primary outcome.
Time Frame: First night after extubation between 11:00pm and 6:00am
Measure: Median (Inter-Quartile Range); unit: miniutes
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 37 | 41
miniutes | 30.5 [16.6 to 64.1] | 16.6 [6.8 to 34.5]

4. Other Pre Specified Outcome: Duration of Sleep During the Day
Description: Continuous EEG-monitoring throughout the day following the sleep trial will be performed until no more than 24 hours after initiation of the sleep trial, or until the patient is discharged from the ICU, whichever occurs first. Duration of sleep during the day will be assessed.
Time Frame: Up to 24 hours after initiation of sleep trial
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 37 | 41
minutes | 553 [507 to 684] | 565.5 [463 to 657]

5. Other Pre Specified Outcome: Subjective Sleep Quality: Richards-Campbell Sleep Questionnaire (RCSQ)
Description: Subjective sleep quality will be assessed by applying the Richards-Campbell Sleep Questionnaire (RCSQ). The RCSQ is a validated survey instrument for assessing sleep quality in critically ill patients based on a five-item, visual analogue scale (each from 0 [worst value] to 100 [best value]). The scale evaluates perceptions of depth of sleep, sleep onset latency, number of awakenings, time spent awake, and overall sleep quality.
Time Frame: Every morning from preoperative day 3 up to postoperative day 7
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 37 | 41
points | 35.47 [24.31 to 46.53] | 34.42 [23.45 to 45.40]

6. Other Pre Specified Outcome: Postoperative Delirium
Description: Incidence of postoperative delirium will be measured daily by the Confusion Assessment Method (CAM) and CAM-ICU. The CAM is a standardized screening tool used for identification of delirium symptoms through a diagnostic algorithm based on 4 cardinal features of delirium, namely acute onset and fluctuating course, inattention, disorganized thinking, and altered level of consciousness. The CAM-ICU, which is routinely performed in the ICU, includes both brief cognitive testing and the CAM algorithm to screen for delirium. For CAM-positive patients, the Delirium Symptom Interview, a standard cognitive assessment consisting of tests of attention, orientation, and memory will be performed by a research team members trained in the survey administration methodology and blinded to treatment assignment to verify the CAM screening results.
Time Frame: Every day from postoperative day 1 up to day of hospital discharge, an expected average of 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 49 | 51
Participants | 10 | 11

7. Other Pre Specified Outcome: Delirium-free Days
Description: as for outcome 6
Time Frame: Every day from postoperative day 1 up to day of hospital discharge, an expected average of 21 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 49 | 51
days | 7 [6 to 10] | 7 [6 to 11]

ADVERSE EVENTS:
Time Frame: from enrollment until discharge
Arm/Group | Suvorexant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 4/49 | 1/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Suvorexant (N=49) | Placebo (N=51)
Somnolence (Nervous system disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Abnormal thought/hallucination (Nervous system disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Metabolic and biochemical derangements in critically ill patients impact drug pharmacokinetics and pharmacodynamics, complicating dose optimization; under the conditions studied, this may have led to an inadequate dose being administered in our study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT04092894/Prot_SAP_000.pdf